CLINICAL TRIAL: NCT00891930
Title: Phase 2 Study of Panitumumab Plus Irinotecan Followed by Panitumumab Plus AMG 479 in Subjects With Metastatic Colorectal Carcinoma Expressing Wild Type KRAS and Refractory to Oxaliplatin-or Irinotecan- and Oxaliplatin-containing Regimens to Evaluate Mechanisms of Acquired Resistance to Panitumumab
Brief Title: Study to Evaluate Mechanisms of Acquired Resistance to Panitumumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NantBioScience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20070820; 2008-004752-77 (EudraCT Number)
Record Dates: First submitted 2009-03-12; First posted 2009-05-01 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2024-07-17 (Actual); Status verified 2024-06

CONDITIONS: Metastatic Colorectal Cancer
Keywords: wild-type KRAS; panitumumab; biomarker; mechanisms of acquired resistance; metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab; ganitumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panitumumab (Experimental): Participants received panitumumab (6 mg/kg starting dose) with irinotecan (starting dose of 180 mg/m²) every 2 weeks (Q2W) during Part 1. Upon radiographically confirmed disease progression, participants proceeded to Part 2 of the study and received treatment with panitumumab (6 mg/kg starting dose) and ganitumab (12 mg/kg starting dose) Q2W.
  Interventions: Biological: Panitumumab; Biological: Ganitumab; Drug: Irinotecan

INTERVENTIONS:
Biological: Panitumumab — Panitumumab 6 mg/kg administered via IV infusion over 60 minutes
  Other Names: Vectibix
Biological: Ganitumab — AMG 479 12 mg/kg adminstered by IV infusion over 60 minutes
  Other Names: AMG 479
Drug: Irinotecan — Irinotecan starting dose of 180 mg/m² adminstered via IV infusion

SUMMARY:
This study is designed to evaluate the mechanism(s) of resistance to the anti-epidermal growth factor receptor (EGFR) antibody panitumumab given in combination with irinotecan in metastatic colorectal carcinoma (mCRC) patients with wild-type Kirsten rat sarcoma-2 virus oncogene (KRAS) tumor status at the time of initial diagnosis.

DETAILED DESCRIPTION:
In Part 1, all participants will undergo a baseline tumor biopsy and will receive panitumumab with irinotecan. Participants who respond or have stable disease will continue to receive treatment until radiographically-confirmed disease progression. These participants will then undergo a second tumor biopsy and blood sampling and then proceed to Part 2 of the study. Participants with radiographically confirmed disease progression at the time of the first tumor measurement will undergo blood sampling and proceed directly to Part 2.

In Part 2, participants will receive panitumumab with ganitumab. In both parts of the study, panitumumab and irinotecan (Part 1) and panitumumab and ganitumab (Part 2) will be administered every 2 weeks until disease progression, intolerability, withdrawal of consent, death, or unless otherwise indicated by the study team.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic adenocarcinoma of the colon or rectum;
* Subjects with wild-type KRAS tumor status confirmed by an Amgen approved central laboratory assessment or an experienced local laboratory assessment of archival tumor tissue (preferably from the primary tumor);
* Radiographic evidence of disease progression while on or ≤ 6 months after completion of treatment with irinotecan- and oxaliplatin- or oxaliplatin-based chemotherapy for mCRC;
* Radiographic measurement of tumor burden done within 28 days prior to Day 1 (start of treatment with investigational product);
* At least 1 uni-dimensionally measurable lesion ≥ 20 mm using conventional computed tomography (CT) or magnetic resonance imaging (MRI) or ≥ 10 mm by spiral CT scan per modified RECIST v1.0. Lesion must not be chosen from a previously irradiated field, unless there has been documented disease progression in that field after irradiation and prior to enrollment. All sites of disease must be evaluated;
* At least 1 tumor (preferably a metastasis or unresected primary tumour) that is amenable to core biopsy, as determined by the clinician who will perform the biopsy;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* A life expectancy estimate of ≥ 3 months;
* Willing to undergo two serial core biopsy procedures of tumors (metastasis or unresected primary);
* other criteria may apply

Exclusion Criteria:

* History of other primary cancer, unless:

  * Malignancy treated with curative intent and with no known active disease present for ≥ 3 years before enrollment and felt to be at low risk for recurrence by the treating physician,
* Adequately treated non-melanomatous skin cancer or lentigo maligna without evidence of disease,

  * Adequately treated cervical carcinoma in situ without evidence of disease,
  * Prostatic intraepithelial neoplasia without evidence of prostate cancer;
* History of prior or concurrent central nervous system (CNS) metastases;
* Prior treatment with anti-EGFR (eg, panitumumab, cetuximab or small molecule inhibitors (eg, erlotinib, gefitinib);
* Prior treatment with monoclonal antibodies directed against insulin-like growth factor-1 receptor (IGF-1R) or small molecule inhibitors directed against IGF-1R;
* Use of systemic chemotherapy or radiotherapy ≤ 21 days before enrollment. Subjects must have recovered from acute toxicities related to radiotherapy;
* Use of any antibody therapy (eg, bevacizumab) ≤ 42 days before enrolment;
* Use of anti-tumor therapies including prior experimental agents or approved anti-tumor small molecules ≤ 30 days before enrolment;
* Known allergy or hypersensitivity to any component of panitumumab, irinotecan, or AMG 479;
* Known uridine diphosphate glucuronosyltransferase 1A1 (UGT1A1) polymorphisms predisposing to increased irinotecan toxicity;
* History of irinotecan intolerance that may interfere with planned treatment;
* History of interstitial lung disease (eg, pneumonitis, pulmonary fibrosis) or evidence of interstitial lung disease on baseline chest CT scan;
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year before enrolment;
* Active inflammatory bowel disease or other active bowel disease causing chronic diarrhea (defined as ≥ grade 2 per Common Terminology Criteria for Adverse Events (CTCAE) version 3.0);
* Known positive test(s) for human immunodeficiency virus (HIV) infection, hepatitis C virus, acute or chronic active hepatitis B infection;
* Major surgical procedure ≤ 28 days before enrollment or minor surgical procedure ≤ 14 days before enrollment. Subjects must have recovered from surgery related toxicities. Core biopsy, central venous catheter placement, fine needle aspiration, thoracentesis, or paracentesis is not considered a major or minor surgical procedure; - Other investigational procedures or drugs (ie, participation in another clinical study) ≤ 30 days before enrolment;
* other criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2009-05-05 (Actual); Primary Completion 2013-07-22 (Actual); Study Completion 2013-07-22 (Actual)

REFERENCES:
- [Derived] Siena S, Sartore-Bianchi A, Garcia-Carbonero R, Karthaus M, Smith D, Tabernero J, Van Cutsem E, Guan X, Boedigheimer M, Ang A, Twomey B, Bach BA, Jung AS, Bardelli A. Dynamic molecular analysis and clinical correlates of tumor evolution within a phase II trial of panitumumab-based therapy in metastatic colorectal cancer. Ann Oncol. 2018 Jan 1;29(1):119-126. doi: 10.1093/annonc/mdx504. PMID 28945848
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Upon radiographically confirmed disease progression per modified RECIST version 1.0, eligible subjects from part 1 proceeded to part 2 of the study to receive panitumumab plus ganitumab.
Groups:
- Overall Study: Period 1:Part 1 Panitumumab + Irinotecan Open label panitumumab 6 mg/kg every 2 weeks plus irinotecan 180 mg/m2 every 2 weeks
  Period 2:Part 2 Panitumumab + AMG479 Treatment with panitumumab 6 mg/kg every 2 weeks plus AMG 479 12 mg/kg every 2 weeks.
Period: Part 1 Panitumumab + Irinotecan
Arm/Group | Overall Study
Started | 74
Completed | 5
Not Completed | 69
Not completed — Full Consent Withdrawn | 2
Not completed — Death | 66
Not completed — Lost to Follow-up | 1
Period: Part 2 Panitumumab + AMG479
Arm/Group | Overall Study
Started | 36 (Subjects that responded (complete or partial response confirmation) or had stable disease (based on modified RECIST v1.0 criteria) continued to receive treatment until radiographically-confirmed disease progression. These subjects proceeded to Part 2 of the study. Subjects that experienced radiographically-confirmed disease progression at the time of first tumor measurement underwent blood sampling then proceeded directly on to Part 2 of the study.)
Completed | 5
Not Completed | 31
Not completed — Full Consent Withdrawn | 1
Not completed — Death | 30

BASELINE CHARACTERISTICS:
Groups:
- Part 1; Part 2: Participants received panitumumab (6 mg/kg starting dose) with irinotecan (starting dose of 180 mg/m²) every 2 weeks (Q2W) during Part 1. Upon radiographically confirmed disease progression, participants proceeded to Part 2 of the study and received treatment with panitumumab (6 mg/kg starting dose) and ganitumab (12 mg/kg starting dose) Q2W.
- Total: Total of all reporting groups
Arm/Group | Part 1 | Part 2 | Total
Number analyzed (Participants) | 74 | 36 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Period 2 part 2 subjects are a subset of period 1 part 1 subjects
  years
    Part 1: number analyzed (Participants) | 74 | 0 | 74
    Part 1 | 62.2 (9.8) |  | 62.2 (9.8)
    Part 2: number analyzed (Participants) | 0 | 36 | 36
    Part 2 |  | 62.9 (10.1) | 62.9 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Period 2 part 2 subjects are a subset of period 1 part 1 subjects
  Participants
    Part 1: number analyzed (Participants) | 74 | 0 | 74
    Part 1: Female | 27 | 0 | 27
    Part 1: Male | 47 | 0 | 47
    Part 2: number analyzed (Participants) | 0 | 36 | 36
    Part 2: Female | 0 | 11 | 11
    Part 2: Male | 0 | 25 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Period 2 part 2 subjects are a subset of period 1 part 1 subjects
  Participants
    Part 1: number analyzed (Participants) | 74 | 0 | 74
    Part 1: American Indian or Alaska Native | 0 | 0 | 0
    Part 1: Asian | 0 | 0 | 0
    Part 1: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Part 1: Black or African American | 0 | 0 | 0
    Part 1: White | 73 | 0 | 73
    Part 1: More than one race | 0 | 0 | 0
    Part 1: Unknown or Not Reported | 1 | 0 | 1
    Part 2: number analyzed (Participants) | 0 | 36 | 36
    Part 2: American Indian or Alaska Native | 0 | 0 | 0
    Part 2: Asian | 0 | 0 | 0
    Part 2: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Part 2: Black or African American | 0 | 0 | 0
    Part 2: White | 0 | 35 | 35
    Part 2: More than one race | 0 | 0 | 0
    Part 2: Unknown or Not Reported | 0 | 1 | 1
Subjects With Metastatic Colorectal Carcinoma Expressing Wild-type KRAS and Refractory to Oxaliplati [Count of Participants; unit: Participants]
  Part 1 | 74 | 0 | 74
  Part 2 | 0 | 36 | 36

OUTCOME MEASURES:

1. Primary Outcome: PFS Hazard Ratio
Description: KRAS mutation status changed from wild-type at baseline to mutant at time of second biopsy in part 1, as measured by the PFS hazard ratio. Hazard ratio is presented as wild-type: mutant
Time Frame: From baseline up to 152 weeks (from baseline to the time of the second biopsy prior to entering part 2) .
Measure: Number (95% Confidence Interval); unit: months
Groups:
- Part 1: Upon radiographically confirmed disease progression, participants proceeded to Part 2 of the study and received treatment with panitumumab (6 mg/kg starting dose) and ganitumab (12 mg/kg starting dose) Q2W.
Arm/Group | Part 1
Number analyzed (Participants) | 74
months | 0.365 [0.164 to 0.808]
Statistical Analysis 1: Comparison: Part 1; Test type: Superiority; p = 0.0130, Regression, Cox

2. Primary Outcome: Objective Response Rate in Part 2
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From time of randomization until confirmed complete response or partial response (part 2: up to 119 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2
Number analyzed (Participants) | 36
percentage of participants | 0.00 [0.00 to 9.74]

3. Secondary Outcome: Objective Response Rate for Part 1
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR.
Time Frame: from first dose of investigational product up to 152 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part 1: Participants received panitumumab (6 mg/kg starting dose) with irinotecan (starting dose of 180 mg/m²) every 2 weeks (Q2W) during Part 1. Upon radiographically confirmed disease progression, participants proceeded to Part 2 of the study and received treatment with panitumumab (6 mg/kg starting dose) and ganitumab (12 mg/kg starting dose) Q2W.
  Panitumumab: Panitumumab 6 mg/kg administered via IV infusion over 60 minutes
Arm/Group | Part 1
Number analyzed (Participants) | 74
percentage of participants | 21.62 [12.89 to 32.72]

4. Secondary Outcome: Progression-Free Survival for Part 1
Description: Time from the first dose of investigational product to the first date of disease progression per the modified RECIST v1.0 or death by any cause, initiating a new line of antitumor therapy, or receiving study treatment in Part 2, whichever is earlier in Part 1. Disease progression is a >= 20% increase in the sum of the longest diameter of the target lesions as compared to the smallest sum while on study per RECIST v1.0
Time Frame: from first dose of investigational product up to 152 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab
Number analyzed (Participants) | 74
months | 4.6 [3.7 to 6.9]

5. Secondary Outcome: Progression-Free Survival for Part 2
Description: Time from the start of Part 2 to the first date of disease progression per the modified RECIST v1.0 or death by any cause, initiating a new line of antitumor therapy, or receiving study treatment in Part 2, whichever is earlier. Disease progression is a >= 20% increase in the sum of the longest diameter of the target lesions as compared to the smallest sum while on study per RECIST v1.0.
Time Frame: 119 weeks from the start of part 2, up to a maximum duration of 152 week
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab
Number analyzed (Participants) | 36
months | 1.7 [1.6 to 1.8]

6. Secondary Outcome: Overall Survival for Part 1
Description: Time from the first dose of investigational product to death from any cause in Part 1.
Time Frame: from first dose of investigational product up to 152 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab
Number analyzed (Participants) | 74
months | 11.6 [7.8 to 12.9]

7. Secondary Outcome: Overall Survival for Part 2
Description: Time from the start of Part 2 to death from any cause.
Time Frame: from the start of Part 2 up to 119 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab
Number analyzed (Participants) | 36
months | 7.6 [5.6 to 12.3]

8. Secondary Outcome: Time to Response for Part 1
Description: Time from the first dose of investigational product to the date of first confirmed objective response in Part 1. An objective response is defined as a confirmed complete response or partial response per modified RECIST v1.0 criteria during the treatment period. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR.
Time Frame: from first dose of investigational product up to 152 weeks
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Panitumumab
Number analyzed (Participants) | 74
months | 2.0 (0.4)

9. Secondary Outcome: Duration of Response for Part 1
Description: Time from first confirmed objective response to disease progression per modified RECIST v1.0 in Part 1. An objective response is defined as a confirmed complete response or partial response per modified RECIST v1.0 criteria during the treatment period. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR; Disease progression is a >= 20% increase in the sum of the longest diameter of the target lesions as compared to the smallest sum while on study.
Time Frame: from first dose of investigational product up to 152 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab
Number analyzed (Participants) | 74
months | 7.7 [6.7 to 9.1]

10. Secondary Outcome: Part 2 Time to Response and Duration of Response
Description: Time to response was defined as the time from study day 1 to the first observation of an objective response (confirmed complete response or partial response using modified Response Evaluation Criteria in Solid Tumors [RECIST]). Duration of response was the time from the first observation of an objective response to the subsequent time of disease progression (per modified RECIST or clinical progression, whichever came first) or death due to any cause. Objective response = a tumor response assessment of either complete response or partial response per modified Response Evaluation Criteria in Solid Tumors [RECIST]. Per RECIST: a complete response is the disappearance of all target lesions; a partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From time of randomization until confirmed complete response or partial response (part 2: up to 119 weeks)
Population: Due to no subjects having complete or partial responses, these Secondary Outcomes were not summarized.
Arm/Group | Part 2
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Part 1: All-Cause Mortality was assessed up to 152 weeks and all other adverse events were collected up to 79 weeks; Part 2: All-Cause Mortality was assessed from start of part 2 up to 119 weeks from time of randomization and all other adverse events were collected up to 41 weeks from time of randomization.
Groups:
- Part 1 Panitumumab + Irinotecan: open label panitumumab 6 mg/kg every 2 weeks plus irinotecan 180 mg/m2 every 2 weeks
- Part 2 Panitumumab + AMG479: treatment with panitumumab 6 mg/kg every 2 weeks plus AMG 479 12 mg/kg every 2 weeks.
Arm/Group | Part 1 Panitumumab + Irinotecan | Part 2 Panitumumab + AMG479
All-Cause Mortality (participants affected / at risk) | 66/74 | 30/36
Serious Adverse Events (participants affected / at risk) | 26/74 | 8/36
Other Adverse Events (participants affected / at risk) | 74/74 | 35/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Panitumumab + Irinotecan (N=74) | Part 2 Panitumumab + AMG479 (N=36)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Asthenia (General disorders) | 3 | 0
Fatigue (General disorders) | 2 | 0
General physical health deterioration (General disorders) | 5 | 2
Performance status decreased (General disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 2 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 1
Anal abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Paresis (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Panitumumab + Irinotecan (N=74) | Part 2 Panitumumab + AMG479 (N=36)
Diarrhoea (Gastrointestinal disorders) | 55 | 8
Asthenia (General disorders) | 41 | 12
Rash (Skin and subcutaneous tissue disorders) | 39 | 15
Nausea (Gastrointestinal disorders) | 38 | 10
Decreased Appetite (Metabolism and nutrition disorders) | 28 | 5
Vomiting (Gastrointestinal disorders) | 28 | 4
Mucosal Inflammation (General disorders) | 25 | 4
Dry Skin (Skin and subcutaneous tissue disorders) | 24 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 23 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 22 | 0
Constipation (Gastrointestinal disorders) | 20 | 8
Skin Fissures (Skin and subcutaneous tissue disorders) | 19 | 3
Abdominal Pain (General disorders) | 18 | 8
Paronychia (Psychiatric disorders) | 18 | 7
Skin Toxicity (Skin and subcutaneous tissue disorders) | 14 | 3
Fatigue (General disorders) | 13 | 5
Pruritus (General disorders) | 13 | 2
Anaemia (Blood and lymphatic system disorders) | 12 | 3
Pyrexia (General disorders) | 12 | 5
Acne (Skin and subcutaneous tissue disorders) | 10 | 2
General Physical Health Deterioration (General disorders) | 10 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 3
Conjunctivitis (Eye disorders) | 9 | 3
Neutropenia (Blood and lymphatic system disorders) | 9 | 2
Weight Decreased (Investigations) | 9 | 0
Abdominal Pain Upper (General disorders) | 8 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 8 | 3
Insomnia (Psychiatric disorders) | 8 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 0
Xerosis (General disorders) | 7 | 2
Dyspepsia (Gastrointestinal disorders) | 6 | 2
Folliculitis (Skin and subcutaneous tissue disorders) | 6 | 2
Headache (General disorders) | 6 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Urinary Tract Infection (Renal and urinary disorders) | 6 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 0
Dysgeusia (Renal and urinary disorders) | 5 | 2
Erythema (General disorders) | 5 | 0
Oedema Peripheral (Nervous system disorders) | 5 | 4
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Paraesthesia (Nervous system disorders) | 5 | 0
Polyneuropathy (Nervous system disorders) | 5 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Stomatitis (Gastrointestinal disorders) | 5 | 2
Trichomegaly (Skin and subcutaneous tissue disorders) | 5 | 0
Abdominal Distension (General disorders) | 4 | 0
Chest Pain (General disorders) | 4 | 0
Dry Eye (Eye disorders) | 4 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Dysuria (Renal and urinary disorders) | 4 | 2
Haematoma (Vascular disorders) | 4 | 0
Haemorrhoids (Vascular disorders) | 4 | 0
Nail Toxicity (Skin and subcutaneous tissue disorders) | 4 | 0
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Neurotoxicity (Nervous system disorders) | 4 | 0
Tachycardia (Cardiac disorders) | 4 | 0
Hypomagnesaemia (General disorders) | 0 | 5
Epistaxis (Ear and labyrinth disorders) | 0 | 3
Infusion Related Reaction (Investigations) | 0 | 3
Nail Bed Inflammation (Skin and subcutaneous tissue disorders) | 0 | 3
Palmar-Plantar Erythrodysaesthesia Syndrome (Nervous system disorders) | 0 | 3
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2
Hepatic Pain (General disorders) | 0 | 2
Hypersensitivity (General disorders) | 0 | 2
Infection (General disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-11-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT00891930/Prot_SAP_000.pdf